CLINICAL TRIAL: NCT01396291
Title: A Double-Blind, Placebo-Controlled Trial of Asenapine in the Prevention of Recurrence of a Mood Episode After Stabilization of an Acute Manic/Mixed Episode in Subjects With Bipolar 1 Disorder (Phase 3B, Protocol P06384)
Brief Title: Efficacy and Safety of Asenapine in the Prevention of Recurrence of Mood Episodes in Participants With Bipolar 1 Disorder (P06384)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06384; 2010-018671-20 (EudraCT Number)
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Bipolar 1 Disorder
MeSH Terms: interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asenapine (Experimental): All study participants will first receive open-label asenapine and placebo for 12 to 16 weeks before being randomized. After randomization, participants will receive asenapine or placebo (this is the double-blind period) for up to 26 weeks.
  Interventions: Drug: asenapine
- Placebo (Placebo Comparator): All study participants will first receive open-label asenapine and placebo for 12 to 16 weeks before being randomized. After randomization, participants will receive asenapine or placebo (this is the double-blind period) for up to 26 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: asenapine — asenapine, sublingual tablets, 5 to 10 mg twice per day (BID)
  Other Names: SCH 900274, Saphris®, Sycrest®, Org 5222
  Arms: Asenapine
Drug: placebo — asenapine-matched placebo, sublingual tablets, BID
  Arms: Placebo

SUMMARY:
This study is being done to evaluate the efficacy and safety of asenapine as compared to placebo in preventing the recurrence of mood episodes after stabilization of an acute/manic mixed episode in participants with Bipolar 1 Disorder. After a Screening Period, each participant will receive open-label asenapine and matching placebo for 12 to 16 weeks. Participants who meet stabilization criteria may then be randomized into one of the two study arms (asenapine or matching placebo) to receive double-blind treatment for up to an additional 26-weeks.

ELIGIBILITY:
Inclusion criteria:

* Male, or a female who is not of child-bearing potential or who is non-pregnant, non-lactating, and is using a medically accepted method of contraception.
* Each participant must be willing and able to provide written informed consent.
* Each participant must have an identified external contact person or an identified responsible person.
* Current diagnosis of Bipolar 1 Disorder, and a current manic (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision [DSM-IV-TR^TM] code 296.4x) or mixed (DSM-IV code 296.6x) episode as determined by a structured clinical interview (Mini International Neuropsychiatric Interview [MINI]) at Screening.
* Each participant must be confirmed to be experiencing an acute manic or mixed bipolar 1 episode.

Exclusion criteria:

* Uncontrolled, unstable clinically significant medical condition.
* Clinically significant abnormal laboratory, vital sign, physical examination, or electrocardiogram findings at Screening.
* Current primary Axis I disorder other than bipolar 1 disorder.
* Meets the current DSM-IV-TR^TM criteria for substance abuse or dependence (excluding nicotine).
* Imminent risk of self-harm or harm to others.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2011-12; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The time (in days) to recurrence of any mood event during the double-blind treatment period | From Week 12 or 16 to Week 38 or 42

CONTACTS AND LOCATIONS:
Locations (80):
- United States (30):
  - Forest Investigative Site 3017, Anaheim, California
  - Forest Investigative Site 3019, Chino, California
  - Forest Investigative Site 3001, Escondido, California
  - Forest Investigative Site 3004, National City, California
  - Forest Investigative Site 3006, Oakland, California
  - Forest Investigative Site 3003, Orange, California
  - Forest Investigative Site 3007, Torrance, California
  - Forest Investigative Site 3042, Colorado Springs, Colorado
  - Forest Investigative Site 3012, Jacksonville, Florida
  - Forest Investigative Site 3040, Kissimmee, Florida
  - Forest Investigative Site 3031, Leesburg, Florida
  - Forest Investigative Site 3015, Miami, Florida
  - Forest Investigative Site 3010, Tampa, Florida
  - Forest Investigative Site 3039, Atlanta, Georgia
  - Forest Investigative Site 3032, Chicago, Illinois
  - Forest Investigative Site 3029, Schaumburg, Illinois
  - Forest Investigative Site 3021, Witchita, Kansas
  - Forest Investigative Site 3014, Gladstone, Missouri
  - Forest Investigative Site 3002, Albuquerque, New Mexico
  - Forest Investigative Site 3024, Elmsford, New York
  - Forest Investigative Site 3037, Avon Lake, Ohio
  - Forest Investigative Site 3041, Cincinnati, Ohio
  - Forest Investigative Site 3023, Oklahoma City, Oklahoma
  - Forest Investigative Site 3035, Oklahoma City, Oklahoma
  - Forest Investigative Site 3033, Memphis, Tennessee
  - Forest Investigative Site 3009, Houston, Texas
  - Forest Investigative Site 3020, Houston, Texas
  - Forest Investigative Site 3036, Irving, Texas
  - Forest Investigative Site 3027, Plano, Texas
  - Forest Investigative Site 3000, Wichita Falls, Texas
- Bulgaria (7):
  - Forest Investigative Site 3105, Pleven, Pleven
  - Forest Investigative Site 3104, Sofia, Sofia-Grad
  - Forest Investigative Site 3100, Sofia, Sofia-Grad
  - Forest Investigative Site 3106, Sofia, Sofia-Grad
  - Forest Investigative Site 3101, Varna, Varna
  - Forest Investigative Site 3102, Burgas
  - Forest Investigative Site 3103, Varna
- Croatia (4):
  - Forest Investigative Site 3153, Zagreb, City of Zagreb
  - Forest Investigative Site 3154, Zagreb, City of Zagreb
  - Forest Investigative Site 3152, Zagreb, City of Zagreb
  - Forest Investigative Site 3156, Rijeka, Rijeka
- India (6):
  - Forest Investigative Site 3308, Nashik, Andhra Pradesh
  - Forest Investigative Site 3306, Ahmedabad, Gujarat
  - Forest Investigative Site 3305, Ahmedabad, Gujaratc
  - Forest Investigative Site 3307, Nashik, Madhya Pradesh
  - Forest Investigative Site 3302, Kanpur, Uttar Pradesh
  - Forest Investigative Site 3303, Hyderabad
- Philippines (4):
  - Forest Investigative Site 3353, Cebu, Cebu
  - Forest Investigative Site 3352, Iloilo City, Iloilo
  - Forest Investigative Site 3356, Mandaluyong, Mandaluyong
  - Forest Investigative Site 3351, Manila, National Capital Region
- Romania (7):
  - Forest Investigative Site 3128, Bucharest, București
  - Forest Investigative Site 3129, Bucharest, București
  - Forest Investigative Site 3130, Bucharest, București
  - Forest Investigative Site 3131, Târgovişte, Dâmbovița County
  - Forest Investigative Site 3125, Iași, Iaşi
  - Forest Investigative Site 3126, Targu Mureş, Mureș County
  - Forest Investigative Site 3127, Arad
- Russia (5):
  - Forest Investigative Site 3205, Kazan', Kazan
  - Forest Investigative Site 3202, Moscow, Moscow
  - Forest Investigative Site 3200, Moscow, Moscow
  - Forest Investigative Site 3201, Saint Petersburg, Sankt-Peterburg
  - Forest Investigative Site 3204, Smolensk, Smolensk Oblast
- Serbia (7):
  - Forest Investigative Site 3177, Belgrade, Belgrade
  - Forest Investigative Site 3176, Belgrade, Beograd
  - Forest Investigative Site 3179, Belgrade, Beograd
  - Forest Investigative Site 3182, Belgrade, Beograd
  - Forest Investigative Site 3178, Kragujevac, Kragujevac
  - Forest Investigative Site 3180, Kragujevac, Kragujevac
  - Forest Investigative Site 3182, Novi Kneževac, Vojvodina
- Turkey (Türkiye) (3):
  - Forest Investigative Site 3252, Korucuk, Adapazari
  - Forest Investigative Site 3255, Ankara, Ankara
  - Forest Investigative Site 3257, Diyarbakır, Diyarbakır
- Ukraine (7):
  - Forest Investigative Site 3230, Chernihiv, Chernihiv Oblast
  - Forest Investigative Site 3228, Kharkiv, Kharkivs’ka Oblast’
  - Forest Investigative Site 3226, Kyiv, Kyiv Oblast
  - Forest Investigative Site 3229, Kyiv, Kyiv Oblast
  - Forest Investigative Site 3227, Luhansk, Luhansk Oblast
  - Forest Investigative Site 3233, Kherson
  - Forest Investigative Site 3232, Lviv

REFERENCES:
- [Derived] Szegedi A, Durgam S, Mackle M, Yu SY, Wu X, Mathews M, Landbloom RP. Randomized, Double-Blind, Placebo-Controlled Trial of Asenapine Maintenance Therapy in Adults With an Acute Manic or Mixed Episode Associated With Bipolar I Disorder. Am J Psychiatry. 2018 Jan 1;175(1):71-79. doi: 10.1176/appi.ajp.2017.16040419. Epub 2017 Sep 26. PMID 28946761